CLINICAL TRIAL: NCT04123717
Title: Pilot Study Comparison Of Intravenous Ibuprofen And Intravenous Paracetamol In Management Of Pediatric Fever
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, DR. KHALID AL-ANSARI, Director of Pediatric Emergency Center's, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 16206/16
Record Dates: First submitted 2019-10-07; First posted 2019-10-11 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Fever
MeSH Terms: conditions — Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm1 - IV Ibuprofen (Active Comparator): Patients will receive IV Ibuprofen 10 mg/kg to a maximum of 400 mg intravenously over 15 minutes. This medication will be diluted as per manufacturer instructions with 100 ml normal saline.
  Interventions: Drug: Intravenous Ibuprofen
- Arm 2 -IV Paracetamol (Active Comparator): Patients will receive 15 mg/kg IV Paracetamol to a maximum of 1000 mg intravenously over 15 minutes. This medication will be diluted as per manufacturer instructions with normal saline.
  Interventions: Drug: Intravenous Ibuprofen
- Arm 3- Both IV Paracetamol and IV Ibuprofen (Active Comparator): Patients will receive an infusion of both IV Paracetamol and IV Ibuprofen. They will initially receive IV Ibuprofen and the IV catheter will then be flushed with 10 ml of normal saline, and the patient will receive IV Paracetamol
  Interventions: Drug: Intravenous Ibuprofen
- Arm 4 -PO Brufen (Active Comparator): Patients will receive PO ibuprofen given as a 100mg/5ml syrup or 200 mg tablets to a maximum of 400 mg. The treating nurse will ask the parental preference to use syrup or tablets. If they vomit the medication within 15 minutes of administration, another full dose will be administered.
  Interventions: Drug: Intravenous Ibuprofen

INTERVENTIONS:
Drug: Intravenous Ibuprofen — The treatment phase consists of assignment to a study arm, either IV Ibuprofen, IV Paracetamol, IV paracetamol-Ibuprofen, or PO ibuprofen, and administration of the appropriate medication. The IV medications will be administered over a 15-minute period. The safety of infusion of IVIbuprofen in just 10 minutes has been established, and to infuse over 15 minutes to ensure that IV Paracetamol and IV Ibuprofen have equal infusion times. For IV paracetamol-Ibuprofen, the IV paracetamol-Ibuprofen will be administered as a sequential infusion of IV Ibuprofen over 15 minutes, followed by a flush of the IV line, followed immediately by IV paracetamol infusion over 15 minutes. Oral ibuprofen will be administered as a syrup or tablet based on patient weight and parental preference.
  Other Names: Intravenous Acetaminophen; Intravenous Acetaminophen & Intravenous Brufen; Brufen PO

SUMMARY:
Fever is one of the most common reasons children are brought to emergency departments. Treatment of fever with antipyretics is usually done simply to make children more comfortable, although in some circumstances, such as febrile seizure, control of fever is critically important.

The investigators seek to compare the two most widely-used IV antipyretic medications, paracetamol and ibuprofen, in multiple measures of fever control. Although there is much data evaluating adults fever, as well as these medications for analgesia in both children and adults, there is scant published data on the topic: One IV Ibuprofen study of 100 children, and one study of IV paracetamol with 67 children.1,6 Due to the highly limited published data evaluating IV ibuprofen and IV paracetamol for pediatric fever due to infection, the investigators seek to conduct a pilot study in order to know the effect size and accurately estimate a sample size in order to design a full randomized controlled trail.

DETAILED DESCRIPTION:
Upon arrival, when patients are found to be febrile, the parent and patient are informed by the treating physician about their study eligibility. They are provided with study information and a consent form, and given the opportunity to discuss the study with a research nurse or assistant.

Within 10 minutes a decision to consent for the study must be made, and if no consent is made the patient is excluded from the study.

After consent into the study, study subjects will be randomized to arm 1,2,3 or 4.

Study Medications: Arm 1,2,3,4:

Will have an intravenous catheter placed by standard method practiced in the Al Saad Pediatric Emergency Center. All febrile patients admitted in the facility have an intravenous catheter placed as a standard practice, so they will not require an IV catheter simply for the purpose of delivering study medications. This will typically be a 24 gauge or 22 gauge angiocatheter, secured with tegaderm and tape. After placement of this IV catheter, the patient will receive the study medication(s).The dosing of these medications, specifically ibuprofen 10 mg/kg and paracetamol 15 mg/kg is standard dosing routinely used in pediatrics.

Arm 1- Patients will receive IV Ibuprofen 10 mg/kg to a maximum of 400 mg intravenously over 15 minutes. This medication will be diluted as per manufacturer instructions with 100 mL normal saline.

Arm 2- Patients will receive 15 mg/kg IV Paracetamol to a maximum of 1000 mg intravenously over 15 minutes. This medication will be diluted as per manufacturer instructions with normal saline.

Arm 3- Patients will receive an infusion of both IV Paracetamol and IV Ibuprofen. They will initially receive IV Ibuprofen as described above. Their IV catheter will then be flushed with 10 ml of normal saline, and the patient will receive IV Paracetamol as described above.

Arm 4- Patients will receive PO ibuprofen given as a 100mg/5ml syrup or 200 mg tablets to a maximum of 400 mg. The treating nurse will ask the parental preference to use syrup or tablets. If they vomit the medication within 15 minutes of administration, another full dose will be administered.

.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 6 months to 14 years.
2. Fever ≥ 38.3°C
3. Admitted to observation unit of Al Saad Pediatric Emergency Center

Exclusion Criteria:

1. Have inadequate intravenous access
2. Have received paracetamol within 4 hours and Ibuprofen within 6 hours before dosing
3. Have fever that is chronic or not new in onset in the preceding 7 days; such as fever from rheumatologic conditions, cancer, or fever of unknown origin, and any fever as a result of transfusion of blood products.
4. Have any history of allergy or hypersensitivity to NSAIDs, aspirin, Paracetamol, or any component of ibuprofen or .Paracetamol
5. Known to have bleeding risk or diathesis such as hemophilia or thrombocytopenia
6. Be receiving ongoing or imminent treatment with corticosteroids
7. Be on dialysis, have oliguria, have impaired renal function or a renal transplant or known renal or hepatic disease
8. Be otherwise unsuitable for the study, in the opinion of the Investigator.
9. Any investigational drug use within 30 days prior to enrollment.

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the Area under the curve for fever in the 4 hours after administration of each study arm relative to Area under the curve for fever of Ibuprofen | 4 hours
  Area under the curve for fever will be calculated as the difference between measured temperature at a given time and 38°C.

SECONDARY OUTCOMES:
Afebrile period/time to first fever recurrence | 6 hours
  Afebrile period as calculated to be the time from first temperature measurement less than 38°C occurring after fever until the first temperature greater than or equal to 38.3°C occurring after fever.

OTHER OUTCOMES:
Febrile seizure occuring within 24 hours of study enrollment | 24 hours
  Safety and tolerability of IV Ibuprofen, IV Paracetamol, IV paracetamol-Ibuprofen, and PO ibuprofen based on Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Alansari, Principal Investigator — Hamad Medical Corporation, Doha, Qatar
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided